CLINICAL TRIAL: NCT01836003
Title: Programmatic CD4 Testing and HAART Initiation Among HIV-Infected Pregnant Women in Gaborone, Botswana: A Randomized Staged Trial of an Improvement Intervention
Brief Title: An Intervention to Improve Antenatal Access to CD4 Testing and HAART in Botswana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Scott Dryden-Peterson, Instructor in Medicine, Harvard Medical School, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BHP044; 3R01HD044391-06S1 (NIH)
Record Dates: First submitted 2013-04-10; First posted 2013-04-19 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: HIV Infection; Pregnancy
Keywords: Pregnancy; Prevention of Mother to Child Transmission; Short Message Service (SMS); HIV infection; CD4 testing; Antiretroviral therapy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tokafatso programmatic intervention (Experimental): Antenatal clinic receives the Tokafatso programmatic intervention, including educational session, SMS-based facilitation of CD4 result delivery, and patient tracing support.
  Interventions: Other: Tokafatso programmatic intervention
- Usual Care (No Intervention): Has not yet received Tokafatso combination programmatic intervention

INTERVENTIONS:
Other: Tokafatso programmatic intervention — Tokafatso programmatic intervention:
  * SMS-based platform for delivery of CD4 test results
  * Participatory educational session for clinic staff
  * Loan program for HIV and CD4 testing supplies
  * Facilitation of tracing of HAART-eligible pregnant women
  Arms: Tokafatso programmatic intervention

SUMMARY:
Access to highly active antiretroviral therapy can improve maternal health outcomes for the 4000 HIV- infected women who give birth daily and nearly eliminate transmission of HIV to their infants. However, system inefficiencies, particularly CD4 testing to determine treatment eligibility, are barriers. The project aims to study the effectiveness of a programmatic intervention at improving antenatal access to treatment.

DETAILED DESCRIPTION:
Perinatal antiretroviral therapy dramatically reduces the risk of transmission of HIV to the 1.4 million infants born annually to HIV-infected mothers. Single-dose and single-drug strategies lead to important reductions in mother-to-child transmission (MTCT). However, more intense strategies using maternal highly active antiretroviral therapy (HAART) to suppress viral replication, lead to 10-fold greater reductions in the risk of MTCT. Wider access to maternal HAART could nearly eliminate the estimated 430,000 annual HIV- infections acquired by infants worldwide. Additionally, prompt initiation of HAART in pregnant women with low CD4+ cell counts could improve maternal mortality and prevent the development of resistant maternal and infant HIV infections.

However, studies from southern Africa, including Botswana, indicate that less than one-third of treatment-eligible women are able to access antenatal HAART. Programmatic inefficiencies in these settings lead to substantial delays in CD4 testing and subsequent treatment initiation. Novel implementation strategies are urgently needed to improve access to the established benefits of antenatal HAART. In collaboration with colleagues in the Botswana Ministry of Health, we have completed an analysis of root causes of the failure to antenatal HAART, identifying delayed CD4 testing and result reporting, and loss-to-follow-up as the principal barriers.

To assess the hypothesis that a low-cost intervention can improve antenatal access to CD4 testing and HAART initiation, the Tokafatso project is a staged-wedge, cluster-randomized study of a combination programmatic intervention. The intervention includes- improved access to CD4 phlebotomy, rapid CD4 result return via SMS messaging, and active follow-up of treatment eligible women. All enrolled clinics will receive the intervention, but the order of implementation will be randomized (10 stages of 2 clinics). Endpoints will be assessed between clinics receiving and not receiving the intervention while adjusting for temporal factors. While clinics will be enrolled and receive the intervention, endpoints will be assessed through anonymous maternity record abstraction of women who subsequently deliver at the catchment inpatient maternity ward.

While tailored to the situation in Botswana, findings are expected to generalizable to implementation of comprehensive prevention of MTCT services throughout the region.

ELIGIBILITY:
Study was conducted and intervention was implemented in antenatal clinics. Criteria for clinic participation:

Inclusion Criteria:

* Clinic providing antenatal services within greater Gaborone, Botswana
* CD4 specimens analyzed at Botswana Harvard HIV Reference Laboratory
* Supervising authority provided written permission for participation

Exclusion Criteria:

* Facilities caring for incarcerated women
* Facilities without a dedicated antenatal program

Endpoints assessed in pregnant women meeting the following criteria:

Inclusion Criteria:

* Delivered at Princess Marina Hospital
* Documented HIV infection
* Botswana citizen

Exclusion Criteria:

* Receiving HAART prior to antenatal clinic registration

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible pregnant women with CD4 enumeration prior to 26 weeks gestation | At delivery
  Gestational age at time of CD4 enumeration will be estimated from last normal menstrual period. Dates of CD4 enumeration and last normal menstrual period will be abstracted from medical records at the time of delivery.
Proportion of eligible women with HAART initiation prior to 30 weeks gestation | At delivery
  Gestational age at time of HAART initiation will be estimated from last normal menstrual period. Dates of HAART initiation and last normal menstrual period will be abstracted from medical records at the time of delivery.

SECONDARY OUTCOMES:
Proportion of eligible women with CD4 testing prior to delivery | At delivery
  Gestational age at time of CD4 enumeration will be estimated from last normal menstrual period. Dates of CD4 enumeration and last normal menstrual period will be abstracted from medical records at the time of delivery.
Proportion of eligible women with HAART initiation prior to delivery | At delivery
  Gestational age at time of HAART initiation will be estimated from last normal menstrual period. Dates of HAART initiation and last normal menstrual period will be abstracted from medical records at the time of delivery.
Gestational age of eligible women at time of CD4 enumeration | At delivery
  Gestational age at time of CD4 enumeration will be estimated from last normal menstrual period. Dates of CD4 enumeration and last normal menstrual period will be abstracted from medical records at the time of delivery.
Gestational age of eligible women at the time of HAART initiation | At delivery
  Gestational age at time of HAART initiation will be estimated from last normal menstrual period. Dates of HAART initiation and last normal menstrual period will be abstracted from medical records at the time of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Dryden-Peterson, MD, Principal Investigator — Harvard School of Public Health, Botswana Harvard AIDS Institute, Brigham and Women's Hospital
Locations (1):
- Botswana Harvard AIDS Institute, Gaborone, Botswana